CLINICAL TRIAL: NCT02567903
Title: Tourniquet Study: Is the High Thrombosis Risk After Knee Arthroscopy Caused by Limb-tourniquet Application? A Randomized Clinical Trial Into the Effect of Tourniquet Use on the Coagulation System
Brief Title: Tourniquet Study: A Clinical Trial Into the Effect of Tourniquet Use on the Coagulation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groene Hart Ziekenhuis (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Ron Onstenk, MD, Groene Hart Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL49117.058.14
Record Dates: First submitted 2015-09-21; First posted 2015-10-05 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Tourniquet (Active Comparator): Knee arthroscopy without the use of a thigh tourniquet.
  Interventions: Procedure: Knee arthroscopy
- Tourniquet (Experimental): Knee arthroscopy with the use of a thigh tourniquet.
  Interventions: Device: Thigh Tourniquet; Procedure: Knee arthroscopy

INTERVENTIONS:
Device: Thigh Tourniquet — Knee arthroscopy with the use of a thigh tourniquet that is inflated to 100-150 mmHg above systolic blood pressure.
  Arms: Tourniquet
Procedure: Knee arthroscopy — Knee arthroscopy

SUMMARY:
Knee arthroscopy is the most commonly performed orthopaedic procedure worldwide, with, according to the American Society for Sports Medicine, over 4 million procedures performed each year. The risk of venous thrombosis following this procedure is considerable with rates of symptomatic events varying between 0.9% and 4.6%. It is currently unknown how this high risk comes about considering its short duration and minimal tissue damage caused by the procedure. A factor that may play a role is the use of a tourniquet. A large majority of orthopaedic surgeons prefer to operate within a 'dry field', which is obtained by the use of a tourniquet. Tourniquet applied surgery is not without risks. Although its use during orthopedic surgery is widely accepted and a standard procedure, tourniquet use can lead to loss of muscle functional strength and contractile speed, vessel wall damage and nerve injury, next to the possibly increased risk of venous thrombosis. In the proposed study the investigators will investigate the effect of a tourniquet on local and systemic markers of hypoxia, inflammation, involvement of endothelium, and coagulation activation. A finding of more prominent activation of the coagulation system with tourniquet use than with non-use will create an important opportunity to prevent thromboembolic events in these patients, as it has been shown that knee arthroscopy can be performed adequately without the use of a tourniquet. Furthermore, it will increase the understanding of the pathophysiology of thrombosis.

DETAILED DESCRIPTION:
Background

Knee arthroscopy is the most commonly performed orthopaedic procedure worldwide, with, according to the American Society for Sports Medicine, over 4 million procedures performed each year. The risk of venous thrombosis following this procedure is considerable with rates of symptomatic events varying between 0.9% and 4.6%.

It is currently unknown how this high risk comes about considering its short duration and minimal tissue damage caused by the procedure. A factor that may play a role is the use of a tourniquet. A large majority of orthopaedic surgeons prefer to operate within a 'dry field', which is obtained by the use of a tourniquet. In the proposed study the investigators will investigate the effect of a tourniquet on local and systemic markers of hypoxia, inflammation, involvement of endothelium, and coagulation activation.

Objective

To investigate the effect of tourniquet application on the coagulation system in patients undergoing a knee arthroscopy. A finding of more prominent activation of the coagulation system with tourniquet use than with non-use will create an important opportunity to prevent thromboembolic events in these patients, as it has been shown that knee arthroscopy can be performed adequately without the use of a tourniquet. Furthermore, it will increase the understanding of the pathophysiology of thrombosis.

Study Design

In a randomized, controlled clinical study the investigators will compare local and systemic coagulation and inflammation markers before and after knee arthroscopy between two groups: 25 patients will be randomized to arthroscopy with tourniquet (Group I) and 25 patients to arthroscopy without tourniquet (Group II).

Inclusion and exclusion criteria

The patients will be recruited from one hospital in Gouda over a 6 months inclusion period. All patients over 18 years, scheduled for a meniscectomy, diagnostic arthroscopy or removal of corpora libera will be eligible for inclusion. Patients will be excluded when they suffer from any kind of coagulation disorder, use of hormonal anticonception, in case of pregnancy or puerperium, when they have a history of venous thrombosis, had major surgery or cast-immobilisation of the lower extremity in the past two months, have a neoplasm or inflammatory disease, have a BMI>30, or when they use anticoagulant therapy. Patients will generally receive spinal anaesthesia. Patients who are nevertheless exposed to any other type of anaesthesia will be excluded as well, to keep the effect of anaesthesia equal for all participants.

Intervention

Patients will be randomized to knee arthroscopy without tourniquet use and to knee arthroscopy with tourniquet use. In patients randomized to arthroscopy with tourniquet use, exsanguination in the leg in which the knee arthroscopy will be performed will be accomplished by raising the leg vertically for one minute. The tourniquet will be inflated to 100-150 mmHg above systolic blood pressure.

Data on duration of surgery and duration of tourniquet use will be collected. Blood collected from the cubital vein and the great saphenous vein during arthroscopy of the knee will be analyzed on outcome parameters that reflect a hypoxic state, an inflammatory reaction, involvement of the endothelium, a procoagulant state and thrombin formation.

Main study endpoints (primary)

Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery will be analyzed.

Different patterns will be analyzed to explore the effect of tourniquet application on the coagulation system by possible biological mechanism. A change (increase or decrease) of markers within one pattern, compared to baseline measurements (before surgery), is considered as a relevant shift of that pattern, thereby suggesting the involvement of that specific pathway.

Outcome parameters that reflect a hypoxic state:

* pH
* pO2
* pCO2
* Lactate

Outcome parameters that reflect an inflammatory reaction:

* White Blood Cell Count (WBCC)
* E-selectin
* Neutrophil Extracellular traps (NETs)

Outcome parameters that reflect involvement of the endothelium:

* Von Willebrand Factor (vWF)
* Thrombomodulin
* E-selectin

Outcome parameters that reflect a procoagulant state and thrombin formation:

* Prothrombin fragments 1+2
* D-dimer
* Plasmin Activator Inhibitor 1 (PAI 1)
* Tissue plasminogen activator (tPA)
* Factor VIII
* Thrombin and Antithrombin complexes (TAT)
* Plasmin and antiplasmin complexes (PAP)

Secondary study paramaters

• Visibility during arthroscopy and technical difficulty score.

Time Schedule

Month 1-3: Completion of study protocol, procedure for approval by METC. Set up of database and randomisation procedure. Instruction of participating clinicians and surgery/anaesthesia staff.

Month 4-6: Inclusion of patients, data collection. Month 7-8: Laboratory tests. Month 9-12: Data analysis, writing and submission of manuscript.

ELIGIBILITY:
Inclusion criteria

* Meniscectomy
* Diagnostic arthroscopy
* Removal of corpora libera

Exclusion Criteria

* Any kind of coagulation disorder
* pregnant or within 3 months of childbirth
* Use of hormonal anticonception
* A history of venous thrombosis
* Had major surgery in the past two months
* A history of cast-immobilization of the lower extremity the past two months
* A neoplasm or inflammatory disease
* A BMI>30
* using anticoagulant therapy
* Any other anaesthesia technique than spinal anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in parameters that reflect a hypoxic state assessed by pH | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in pH between timepoints
Change in parameters that reflect a hypoxic state assessed by pO2 | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in pO2 between timepoints
Change in parameters that reflect a hypoxic state assessed by pCO2 | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in pCO2 between timepoints
Change in parameters that reflect a hypoxic state assessed by Lactate | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Lactate between timepoints
Change in parameters that reflect an inflammatory reaction assessed by WBCC | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in White Blood Cell Count (WBCC) between timepoints
Change in parameters that reflect an inflammatory reaction and/or endothelium involvement assessed by E-selectin | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in E-selectin between timepoints
Change in parameters that reflect an inflammatory reaction assessed by NETs | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Neutrophil Extracellular traps (NETs) between timepoints
Outcome parameters that reflect involvement of the endothelium assessed by vWF | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Von Willebrand Factor (vWF) between timepoints
Outcome parameters that reflect involvement of the endothelium assessed by thrombomodulin. | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Thrombomodulin between timepoints
Outcome parameters that reflect involvement of the endothelium assessed by f 1+2 | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Prothrombin fragments 1+2 (f 1+2) between timepoints
Outcome parameters that reflect a procoagulant state and thrombin formation assessed by D-dimer | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in D-dimer between timepoints
Outcome parameters that reflect a procoagulant state and thrombin formation assessed by PAI 1 | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Plasmin Activator Inhibitor 1 (PAI 1) between timepoints
Outcome parameters that reflect a procoagulant state and thrombin formation assessed by tPA | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Tissue plasminogen activator (tPA) between timepoints
Outcome parameters that reflect a procoagulant state and thrombin formation assessed by factor VIII | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Factor VIII between timepoints
Outcome parameters that reflect a procoagulant state and thrombin formation assessed by TAT | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Thrombin and Antithrombin complexes (TAT) between timepoints
Outcome parameters that reflect a procoagulant state and thrombin formation assessed by PAP | Change in parameters between timepoints; Before surgery (blood drawn approximately 1 hour before surgery), directly after surgery (blood drawn within 5 minutes), 1 hour after surgery.
  Change in Plasmin and antiplasmin complexes (PAP) between timepoints

SECONDARY OUTCOMES:
Duration of surgery | intraoperative, duration in minutes between first incision until closure
  The total duration of surgery in minutes
Duration of tourniquet use | intraoperative, duration in minutes between tourniquet inflation and deflation
  The total duration of tourniquet inflation in minutes
Per-operative visibility | Per-operative
  Visibility during surgery, measured on a Visual Analogue Scale scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C Cannegieter, MD, PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Groene Hart Ziekenhuis, Gouda, South Holland, Netherlands

REFERENCES:
- [Background] American Academy of Orthopaedic Surgeons. Knee Arthroscopy. 2013. http://orthoinfo.aaos.org/topic.cfm?topic=a00299. Accessed April 15, 2014
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Hoppener MR, Ettema HB, Kraaijenhagen RA, Verheyen CC, Henny PC. Day-care or short-stay surgery and venous thromboembolism. J Thromb Haemost. 2003 Apr;1(4):863-5. doi: 10.1046/j.1538-7836.2003.t01-9-00115.x. No abstract available. PMID 12871434
- [Background] Hoppener MR, Ettema HB, Henny CP, Verheyen CC, Buller HB. Symptomatic deep vein thrombosis and immobilization after day-care arthroscopy of the knee. J Thromb Haemost. 2005 Jan;3(1):185-7. doi: 10.1111/j.1538-7836.2004.01091.x. No abstract available. PMID 15634289
- [Background] Hoppener MR, Ettema HB, Henny CP, Verheyen CC, Buller HR. Low incidence of deep vein thrombosis after knee arthroscopy without thromboprophylaxis: a prospective cohort study of 335 patients. Acta Orthop. 2006 Oct;77(5):767-71. doi: 10.1080/17453670610012962. PMID 17068708
- [Background] Camporese G, Bernardi E, Prandoni P, Noventa F, Verlato F, Simioni P, Ntita K, Salmistraro G, Frangos C, Rossi F, Cordova R, Franz F, Zucchetta P, Kontothanassis D, Andreozzi GM; KANT (Knee Arthroscopy Nadroparin Thromboprophylaxis) Study Group. Low-molecular-weight heparin versus compression stockings for thromboprophylaxis after knee arthroscopy: a randomized trial. Ann Intern Med. 2008 Jul 15;149(2):73-82. doi: 10.7326/0003-4819-149-2-200807150-00003. PMID 18626046
- [Background] Ilahi OA, Reddy J, Ahmad I. Deep venous thrombosis after knee arthroscopy: a meta-analysis. Arthroscopy. 2005 Jun;21(6):727-30. doi: 10.1016/j.arthro.2005.03.007. PMID 15944631
- [Background] Ramos J, Perrotta C, Badariotti G, Berenstein G. Interventions for preventing venous thromboembolism in adults undergoing knee arthroscopy. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD005259. doi: 10.1002/14651858.CD005259.pub3. PMID 18843687
- [Background] Bovill EG, van der Vliet A. Venous valvular stasis-associated hypoxia and thrombosis: what is the link? Annu Rev Physiol. 2011;73:527-45. doi: 10.1146/annurev-physiol-012110-142305. PMID 21034220
- [Background] Aglietti P, Baldini A, Vena LM, Abbate R, Fedi S, Falciani M. Effect of tourniquet use on activation of coagulation in total knee replacement. Clin Orthop Relat Res. 2000 Feb;(371):169-77. doi: 10.1097/00003086-200002000-00021. PMID 10693564
- [Background] Katsumata S, Nagashima M, Kato K, Tachihara A, Wauke K, Saito S, Jin E, Kawanami O, Ogawa R, Yoshino S. Changes in coagulation-fibrinolysis marker and neutrophil elastase following the use of tourniquet during total knee arthroplasty and the influence of neutrophil elastase on thromboembolism. Acta Anaesthesiol Scand. 2005 Apr;49(4):510-6. doi: 10.1111/j.1399-6576.2005.00621.x. PMID 15777299
- [Background] Kageyama K, Nakajima Y, Shibasaki M, Hashimoto S, Mizobe T. Increased platelet, leukocyte, and endothelial cell activity are associated with increased coagulability in patients after total knee arthroplasty. J Thromb Haemost. 2007 Apr;5(4):738-45. doi: 10.1111/j.1538-7836.2007.02443.x. PMID 17408407
- [Background] Reikeras O, Clementsen T. Time course of thrombosis and fibrinolysis in total knee arthroplasty with tourniquet application. Local versus systemic activations. J Thromb Thrombolysis. 2009 Nov;28(4):425-8. doi: 10.1007/s11239-008-0299-6. Epub 2008 Dec 6. PMID 19067121
- [Background] Sharrock NE, Go G, Sculco TP, Ranawat CS, Maynard MJ, Harpel PC. Changes in circulatory indices of thrombosis and fibrinolysis during total knee arthroplasty performed under tourniquet. J Arthroplasty. 1995 Aug;10(4):523-8. doi: 10.1016/s0883-5403(05)80155-x. PMID 8523013
- [Background] Estebe JP, Davies JM, Richebe P. The pneumatic tourniquet: mechanical, ischaemia-reperfusion and systemic effects. Eur J Anaesthesiol. 2011 Jun;28(6):404-11. doi: 10.1097/EJA.0b013e328346d5a9. PMID 21502865
- [Background] Johnson DS, Stewart H, Hirst P, Harper NJ. Is tourniquet use necessary for knee arthroscopy? Arthroscopy. 2000 Sep;16(6):648-51. doi: 10.1053/jars.2000.4826. PMID 10976127
- [Background] Kam PC, Kavanagh R, Yoong FF. The arterial tourniquet: pathophysiological consequences and anaesthetic implications. Anaesthesia. 2001 Jun;56(6):534-45. doi: 10.1046/j.1365-2044.2001.01982.x. PMID 11412159
- [Background] Alcelik I, Pollock RD, Sukeik M, Bettany-Saltikov J, Armstrong PM, Fismer P. A comparison of outcomes with and without a tourniquet in total knee arthroplasty: a systematic review and meta-analysis of randomized controlled trials. J Arthroplasty. 2012 Mar;27(3):331-40. doi: 10.1016/j.arth.2011.04.046. Epub 2011 Sep 22. PMID 21944371
- [Background] Hoogeslag RA, Brouwer RW, van Raay JJ. The value of tourniquet use for visibility during arthroscopy of the knee: a double-blind, randomized controlled trial. Arthroscopy. 2010 Sep;26(9 Suppl):S67-72. doi: 10.1016/j.arthro.2009.12.008. Epub 2010 May 13. PMID 20810094
- [Background] Schreijer AJ, Cannegieter SC, Meijers JC, Middeldorp S, Buller HR, Rosendaal FR. Activation of coagulation system during air travel: a crossover study. Lancet. 2006 Mar 11;367(9513):832-8. doi: 10.1016/S0140-6736(06)68339-6. PMID 16530577